CLINICAL TRIAL: NCT01121848
Title: A Randomized Phase III Study of 5-Fluorouracil-based Regimen With or Without Oxaliplatin as 2nd Line Treatment of Advanced or Metastatic Pancreatic Cancer in Patients Who Have Previously Received Gemcitabine-based Chemotherapy
Brief Title: Randomized Study With Oxaliplatin in 2nd Line Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OXALI_L_04918; U1111-1116-9746 (Other: UTN)
Record Dates: First submitted 2010-04-29; First posted 2010-05-12 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Leucovorin; Oxaliplatin; Fluorouracil

ARMS (2):
- 5-FU & LV (Active Comparator): * Day 1: LV 400 mg/m2 (given as a 2-hour infusion)
  * Day 1 and 2: 5-FU given as a bolus IV 400 mg/m2 dose on Day 1 followed by 2400 mg/m2 continuous infusion over 46 hours.
  * This chemotherapy regimen will be administered each two weeks.
  Interventions: Drug: Leucovorin; Drug: 5-Fluorouracil
- XELOX or modified FOLFOX-6 (Experimental): XELOX:
  * Day 1: Oxaliplatin 130 mg/m2 (2 hours infusion)
  * This chemotherapy regimen will be administered each two weeks.
  OR modified FOLFOX-6:
  * Day 1: Oxaliplatin 85 mg/m2 (given as a 2-hour infusion)
  * Day 1: LV 400 mg/m2 (given as a 2-hour infusion simultaneous to oxaliplatin)
  * Day 1 and 2: 5-FU given as a bolus IV 400 mg/m2 dose on Day 1 followed by 2400 mg/m2 continuous infusion over 46 hours (Day 1 and 2)
  * This chemotherapy regimen will be administered each two weeks.
  Interventions: Drug: Leucovorin; Drug: OXALIPLATIN; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Leucovorin — Pharmaceutical form:vials of 50 mg/5 mL or 500 mg/50mL Route of administration: IV
  Dose regimen:
Drug: OXALIPLATIN — Pharmaceutical form: Lyophilized powder for injection (50 mg/vial or 100 mg/vial) or aqueous solution (50 mg/10 mL and 100 mg/20 mL) Route of administration: IV
  Dose regimen:
  Arms: XELOX or modified FOLFOX-6
Drug: 5-Fluorouracil — Pharmaceutical form: vials of 5 g/100mL Route of administration: IV
  Dose regimen:

SUMMARY:
Primary Objective:

To demonstrate that the addition of oxaliplatin to 5-Fluorouracil (5-FU) and Leucovorin (LV) will improve the Progression-Free Survival (PFS). Progression is based on RECIST (Response Evaluation Criteria In Solid Tumors) criteria or death

Secondary Objective:

To evaluate other measures of tumor responses, safety, quality of life (QoL), and health utility assessment.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically proven pancreatic carcinoma
* Measurable locally advanced or metastatic disease
* Patient previously treated with 5-FU as a "radiation sensitizer" and all toxicities must have been resolved
* Patients must have received Gemcitabine-based chemotherapy (single agent or combination) as 1st line therapy for advanced or metastatic disease and all toxicities must have been resolved
* Patients received the last dose of gemcitabine at least 2 weeks prior to randomization
* Confirmed radiographic disease progression (Computed Tomogram (CT) scan or Magnetic Resonance Imaging (MRI) within 4 weeks prior to randomization
* Adequate liver and kidney function:

  * Total bilirubin inferior than 1.5 Upper Limit of Normal (ULN)
  * Creatinine clearance (ClCr) superior than 50 mL / min
  * Aspartate Transferase (AST) inferior than 3 ULN if no liver metastasis or AST inferior than 5 ULN if liver metastasis
  * Alanine Aminotransferase (ALT) inferior than 3 ULN if no liver metastasis or ALT inferior than 5 ULN if liver metastasis
* Adequate hematological function:

  * Neutrophils superior or egal to 1.5 x 109/L
  * Platelets superior or egal to 100 x 109/L

Exclusion criteria:

* Peripheral sensory or motor neuropathy > grade 1
* Eastern Cooperative Oncology Group (ECOG) Performance status > 2
* Serious cardiac arrhythmia, diabetes, or serious active infection or other active illness that would preclude study participation in the opinion of the investigator
* Pernicious anemia or other megaloblastic anemia with vitamin B12 deficiency
* Previous (greater than 5 years) or current malignancies of other origin within the past 5 years
* Lack of physical integrity of the upper gastrointestinal tract, clinically significant malabsorption syndrome, or inability to take oral medications
* History of known allergy to oxaliplatin or other platinum compounds, to 5-FU, to LV or to any ingredients in the formulations or the containers
* Severe renal impairment (ClCr < 50 mL/min)
* Pregnant women or breast-feeding
* Patients (male or female) with reproductive potential not implementing accepted and effective method of contraception (the definition of "effective method of contraception" will be based on the investigators' judgment)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Within the 3 months of study treatment
  PFS is defined as the time from the start of treatment to the date of disease progression or death from any cause.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 12 weeks
  ORR is based on RECIST criteria and is the percentage of patients with complete response (CR) or partial response (PR).
Duration of response | 12 weeks
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever status is recorded first) until the first date that recurrence, i.e. progressive disease (PD) is determined by RECIST criteria or death
Disease Controlled Rate (DCR) | 12 weeks
  DCR is also based on RECIST criteria and is defined as the percentage of patients who have a CR, PR or stable disease (SD)
Median Overall Survival (OS) | 2 years
  Median Survival is the number of weeks at which 50% of the patients are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (15):
- Canada (15):
  - Investigational Site Number 124015, Abbotsford
  - Investigational Site Number 124018, Brampton
  - Investigational Site Number 124014, Burnaby
  - Investigational Site Number 124006, Calgary
  - Investigational Site Number 124008, Greater Sudbury
  - Investigational Site Number 124011, Greenfield Park
  - Investigational Site Number 124010, Hamilton
  - Investigational Site Number 124-016, New Glasgow
  - Investigational Site Number 124013, Oshawa
  - Investigational Site Number 124012, Ottawa
  - Investigational Site Number 124004, Sherbrooke
  - Investigational Site Number 124007, Surrey
  - Investigational Site Number 124003, Toronto
  - Investigational Site Number 124002, Toronto
  - Investigational Site Number 124001, Vancouver

REFERENCES:
- [Derived] Gill S, Ko YJ, Cripps C, Beaudoin A, Dhesy-Thind S, Zulfiqar M, Zalewski P, Do T, Cano P, Lam WYH, Dowden S, Grassin H, Stewart J, Moore M. PANCREOX: A Randomized Phase III Study of Fluorouracil/Leucovorin With or Without Oxaliplatin for Second-Line Advanced Pancreatic Cancer in Patients Who Have Received Gemcitabine-Based Chemotherapy. J Clin Oncol. 2016 Nov 10;34(32):3914-3920. doi: 10.1200/JCO.2016.68.5776. Epub 2016 Sep 30. PMID 27621395